CLINICAL TRIAL: NCT00905970
Title: Demonstration of the Dynamic Hypothesis of Latent Tuberculosis Infection
Acronym: HYPDYN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other)
Responsible Party: Dr. Pere-Joan Cardona, Experimental Tuberculosis Unit. Fundació Institut Germans Trias i Pujol
Other Study IDs: HYPDYN; CEIC EO-07-033
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Last update posted 2011-07-11 (Estimated); Status verified 2009-11

CONDITIONS: Latent Tuberculosis Infection
MeSH Terms: conditions — Latent Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood collected on QuantiFeron-Gold-In Tube tubes. Exhaled breath collected on R-Tube
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- 1: Patients with LTBI recently diagnosed under prophylactic chemotherapy treatment.
- 2: Patients with LTBI recently diagnosed not following any prophylactic chemotherapy treatment.
- 3: Patients with LTBI diagnosed time ago.
- 4: Positive control for the Exhaled Breath condensate assay only. Patients with active TB will conform this group. The n of this group is determined, as it will only be used as a positive control to prove the bacilli's DNA can be detected in the exhaled breath condensate.

SUMMARY:
It is traditionally considered that the development of Latent Tuberculosis Infection (LTBI) is due to the M. tuberculosis ability to develop a dormancy state within well-structured lesions (granulomas), which can remain in the lung of the host even for life. A new original hypothesis has been developed in the Experimental Tuberculosis Unit based on scientific evidence that take into account the idea that a lesion cannot be held forever, because the host tends to remove any lesion in order to rebuild the original parenchyma, in a healing process. Even if M. tuberculosis can remain in a dormant/non-replicating state for a long period, this is an important but not sufficient factor to explain the LTBI. The Dynamic Hypothesis tries to explain the existence of LTBI in spite of the healing process that could remove it by a constant reinfection of the host's tissue. While the "Static" view defends the induction of active TB after the reactivation of the bacilli from and old lesion; while the "Dynamic" view wants to demonstrate that there is a constant induction of new granulomas. In case one of these new lesions takes place in the upper lobe privileged zone, the possibility to induce a cavity would appear, developing an active Tuberculosis (TB).

ELIGIBILITY:
Inclusion Criteria:

* being at least 18 years old
* to be M.tuberculosis infected (diagnosed by a positive TST with or without a positive result in the QuantiFeron-TB-Gold In tube assay)

Exclusion Criteria:

* active TB
* individuals not willing to participate in the study and or not willing to sign the informed consent form
* individuals not able to decide their participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Latent Tuberculosis Infected people
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2009-05; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
QuantiFeron-Gold-In Tube method assay | Every 6 months during 3 years
Detection of M.tuberculosis DNA and RNA in the exhaled breath condensate | Once every year (every 6 months if possible), during 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Pere-Joan Cardona, MD, PhD, Principal Investigator — Fundació Institut Germans Trias i Pujol
Locations (1):
- Fundació Institut Germans Trias i Pujol, Badalona, Barcelona, Spain

REFERENCES:
- [Background] Cardona PJ. A dynamic reinfection hypothesis of latent tuberculosis infection. Infection. 2009 Apr;37(2):80-6. doi: 10.1007/s15010-008-8087-y. Epub 2009 Mar 23. PMID 19308318
- [Background] Caceres N, Tapia G, Ojanguren I, Altare F, Gil O, Pinto S, Vilaplana C, Cardona PJ. Evolution of foamy macrophages in the pulmonary granulomas of experimental tuberculosis models. Tuberculosis (Edinb). 2009 Mar;89(2):175-82. doi: 10.1016/j.tube.2008.11.001. Epub 2008 Dec 24. PMID 19110471
- [Background] Cardona PJ. New insights on the nature of latent tuberculosis infection and its treatment. Inflamm Allergy Drug Targets. 2007 Mar;6(1):27-39. doi: 10.2174/187152807780077282. PMID 17352686
- [Background] Mack U, Migliori GB, Sester M, Rieder HL, Ehlers S, Goletti D, Bossink A, Magdorf K, Holscher C, Kampmann B, Arend SM, Detjen A, Bothamley G, Zellweger JP, Milburn H, Diel R, Ravn P, Cobelens F, Cardona PJ, Kan B, Solovic I, Duarte R, Cirillo DM; C. Lange; TBNET. LTBI: latent tuberculosis infection or lasting immune responses to M. tuberculosis? A TBNET consensus statement. Eur Respir J. 2009 May;33(5):956-73. doi: 10.1183/09031936.00120908. PMID 19407047